CLINICAL TRIAL: NCT04202328
Title: A Retrospective Study for Evaluation of Real-world Efficacy and Safety of T-DM1 in HER2-positive Locally-advanced Unresectable or Metastatic Breast Cancer
Brief Title: T-DM1 in HER2-positive Metastatic/Relapsed Breast Cancer
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Samsung Medical Center (Other)
Collaborators: Health Insurance Review & Assessment Service (Unknown); Korean Cancer Study Group (Other)
Responsible Party: Principal Investigator, Yeon Hee Park, Professor, Samsung Medical Center
Other Study IDs: KCSG BR19-15
Record Dates: First submitted 2019-12-09; First posted 2019-12-17 (Actual); Last update posted 2019-12-19 (Actual); Status verified 2019-12

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a retrospective, multicenter, non-interventional study for the evaluation of real-world efficacy and safety of T-DM1 in metastatic/relapsed HER2-positive breast cancer as part of the establishment of hospital medical record collection system to evaluate drug effectiveness by Health Insurance Review & Assessment Service (HIRA). The medical records in approximately 1,000 patients of HER2-positive locally-advanced unresectable or metastatic breast cancer, who have received Kadcyla(Trastuzumab Emtansine, T-DM1) previously, will be collected.

DETAILED DESCRIPTION:
T-DM1 therapy has shown a survival benefit in previously trastuzumab-treated HER2-positive locally-advanced unresectable or metastatic breast cancer patients from clinical trials. However, the real-world efficacy and safety of T-DM1 in KOREA were not evaluated outside the controlled clinical trials. Therefore, this large multicenter retrospective analysis was designed to evaluate the real-world efficacy and safety of T-DM1 under the Korea National Health Insurance System. The medical records in approximately 1,000 patients with relapsed or De Novo metastatic breast cancer, who have received T-DM1 between Aug 03, 2017 and Dec 31, 2018 will be collected. Eligibility criteria included age ≥ 19 years, histologically confirmed HER2-positive, relapsed after primary surgery or initially metastatic breast cancer, and previous trastuzumab treated. Efficacy was evaluated by overall survival, progression free survival, time to progression, objective response rate, disease control rate, duration of response and time to next treatment. Safety was evaluated by hematologic or non-non hematologic toxicities and adverse events of special interest with T-DM1 therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥19 years at the time of study registration
2. Participants must have histologically confirmed HER2-positive breast cancer
3. Locally advanced unresectable or metastatic patients
4. Patients who have received T-DM1 therapy between Aug 2017 and December 2018 under the Korea National Health Insurance System

Exclusion Criteria:

• Patients who have received T-DM1 therapy outside of the Korea National Health Insurance System

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients with locally-advanced unresectable or metastatic HER2-positive breast cancer, who have received T-DM1 therapy between Aug 2017 and December 2018 under the Korea National Health Insurance System
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-19 (Estimated); Primary Completion 2020-07-31 (Estimated); Study Completion 2020-07-31 (Estimated)

PRIMARY OUTCOMES:
Progression free Survival, PFS | Until September 30, 2019
  Time from the start of T-DM1 to disease progression or death from any cause
Incidence of adverse events | Until September 30, 2019
  Number (percentage) of subjects reporting adverse events

SECONDARY OUTCOMES:
Time to Next Treatment, TTNT | Until September 30, 2019
  Time from the end of T-DM1 to institution of next systemic therapy
Objective Response Rate, ORR | Until September 30, 2019
  The proportion of subjects confirmed complete or partial response
Overall Survival, OS | Until September 30, 2019
  Time from the start of T-DM1 to death from any cause
Disease Control Rate, DCR | Until September 30, 2019
  The proportion of subjects confirmed complete or partial response or stable disease
Duration of response | Until September 30, 2019
  Time from documentation of tumor response to disease progression
Adverse events of special interest | Until September 30, 2019
  Number (percentage) of subjects reporting adverse events of special interest associated with T-DM1

CONTACTS AND LOCATIONS:
Locations (60):
- South Korea (60):
  - Korea University Ansan Hospital, Ansan
  - Hallym University Sacred Heart Hospital, Anyang
  - Soonchunhyang University Bucheon Hospital, Bucheon-si
  - The Catholic University of Korea, Bucheon ST. Mary's Hospital, Bucheon-si
  - Dongnam Institute of Radiological&Medical Sciences, Busan
  - Inje University Busan Paik Hospital, Busan
  - Dong-A University Hospital, Busan
  - Pusan National University Hospital, Busan
  - Kosin University Gospel Hospital, Busan
  - Gyeongsang National University Changwon Hospital, Changwon
  - Dankook University Hospital, Cheonan
  - Soonchunhyang University Cheonan Hospital, Cheonan
  - Chungbuk National University Hospital, Cheonju
  - Daegu Fatima Hospital., Daegu
  - Kyungpook National University Chilgok Hospital, Daegu
  - Yeungnam University Medical Center, Daegu
  - Daegu Catholic University Medical Center, Daegu
  - Keimyung University Dongsan Medical Center, Daegu
  - The Catholic University of Korea Daejeon ST. Mary's Hospital, Daejeon
  - Chungnam National University Hospital, Daejeon
  - Daejeon Eulji Medical Center, Eulji University., Daejeon
  - Konyang University Hospital, Daejeon
  - Gangneung Asan Hospital, Gangneung
  - National Cancer Center, Goyang
  - Chosun University Hospital, Gwangju
  - Dongguk University Gyeongju Hospital., Gyeongju
  - Hallym University Dongtan Sacred Heart Hospital, Hwaseong-si
  - Chonnam National University Hwasun Hospital, Hwasun
  - Dongguk University Ilsan Hospital, Ilsan
  - nje University Ilsan Paik Hospital, Ilsan
  - The Catholic University of Korea Incheon ST. Mary's Hospital, Incheon
  - Gachon University Gil Medical Center, Incheon
  - Inha University Hospital, Incheon
  - Chonbuk National University Hospital, Jeonju
  - Gyeongsang National University Hospital, Jinju
  - Cha University Bundang Medical Center, Seongnam
  - Seoul National University Bundang Hospital, Seongnam
  - Korea Cancer Hospital of Korea Institute of Radiological and Medical Sciences, Seoul
  - Nowon Eulji Medical Center, Eulji University, Seoul
  - Kangdong Kyung Hee University Medical Center, Seoul
  - Korea University Anam Hospital, Seoul
  - Seoul National University Hospital, Seoul
  - Kangbuk Samsung Hospital, Seoul
  - Severance Hospital, Yonsei University Health System, Seoul
  - Soonchunhyang University Seoul Hospital, Seoul
  - Konkuk University Medical Center, Seoul
  - Asan Medical Center, Seoul
  - Gangnam Severance Hospital, Seoul
  - Samsung Medical Center, Seoul
  - The Catholic University of Korea Seoul ST. Mary's Hospital, Seoul
  - ChungAng University Hospital, Seoul
  - SMG-SNU Boramae Medical Center, Seoul
  - The Catholic University of Korea Yeouido ST. Mary's Hospital, Seoul
  - Hallym University Kangnam Sacred Heart Hospital, Seoul
  - Ewha Womans University Mokdong Hospital, Seoul
  - The Catholic University of Korea ST. Mary's Hospital, Suwon
  - Ajou University Hospital, Suwon
  - The Catholic University of Korea Uijeongbu ST. Mary's Hospital, Uijeongbu-si
  - Ulsan University Hospital, Ulsan
  - Pusan National University Yangsan Hospital, Yangsan